CLINICAL TRIAL: NCT02987309
Title: Indirect Calorimetry: SensorMedics Vmax vs GE Carescape - a Method Comparison Study
Status: Terminated | Type: Observational
Why Stopped: Equipment failure
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Gunnar Bentsen, Principal Investigator, Oslo University Hospital
Other Study IDs: 2016_InKal1
Record Dates: First submitted 2016-11-18; First posted 2016-12-08 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Nutrition Assessment; Critical Illness; Children
Keywords: indirect calorimetry; method comparison
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Dosing of nutrition in PICUs is mainly based on patient weight and assumptions on clinical status. There is however poor correlation between these calculations and actual energy consumption measured with indirect calorimetry (IC). Available equipment for IC has however been too cumbersome to use in daily clinical practice. Of relative new date is IC integrated in modern ventilators. This functionality is easy to use, but we do not know if the results are reliable for children. This study is a method comparison study comparing measurements done with SensorMedics Vmax ("gold standard") vs GE Carescape (modern ventilator with Integrated IC) in children undergoing intensive care treatment.

ELIGIBILITY:
Inclusion Criteria:

* < 18 years of age,
* endotracheally intubated.
* FiO2 < 0,6, tube leak < 10%, tidal volume > 50 ml.

Exclusion Criteria:

* Ventilatory and hemodynamically unstable during 2 hours prior to inclusion.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children undergoing intensive care treatment
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
MEE (measured energy expenditure) kcal/kg/day, RQ (respiratory quotient) | 2 hours
  Comparison of measurements made by two different instruments

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Bentsen, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No